CLINICAL TRIAL: NCT03700827
Title: Effects of Aerobic and Resistance Training on Abdominal Fat Loss
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Southern Illinois University Edwardsville (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-1208-4C-2
Record Dates: First submitted 2018-09-05; First posted 2018-10-09 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-03

CONDITIONS: Obesity, Abdominal
Keywords: Abdominal Fat; Visceral Adipose Tissue; Subcutaneous Adipose Tissue; Exercise; Intervention
MeSH Terms: conditions — Obesity, Abdominal; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resistance Training Group (Experimental): Resistance training will consist of 3 whole body circuits per week for 3 weeks lasting approximately 1 hour per session. All major muscle groups will be involved (leg press, bent-over-row, bench press, back squat, dumbbell jump squats, dead-lifts, and weighted abdominal crunches). Each participant will go through each circuit three times with 30 seconds between each exercise and 2 minutes between each set.
  Interventions: Other: Resistance Training
- Aerobic Training Group (Experimental): Aerobic interval training will consist of 3 sessions/week for 3 weeks for approximately 45-50 minutes per session depending on exercise energy expenditure. There will be two periods of intervals. The first period will be 3 minutes of high-intensity activity and the second period will be reduced to moderate-intensity for 2 minutes. The speed/incline will change depending on the participants perception or Borg's rating of perceived exertion. Intensity will be measured using Lactate levels after each session.
  Interventions: Other: Aerobic Training
- Control Group (No Intervention): The control group must attend sessions but will not exercise.

INTERVENTIONS:
Other: Resistance Training — High-intensity Resistance Training Group
  Arms: Resistance Training Group
Other: Aerobic Training — Aerobic Interval Training Group
  Arms: Aerobic Training Group

SUMMARY:
Study the effects of different exercise modes on total and regional adiposity variation in subcutaneous and visceral adipose tissue (VAT and SAT). The investigators hypothesize that total abdominal will improve for all the exercise groups compared to the control group. When comparing intervention groups: 1) no differences on the degree of improvement in total abdominal fat depots (VAT and SAT) 2) different degree of change when comparing specific sections at VAT and SAT are expected.

ELIGIBILITY:
Inclusion Criteria:

* 30 - 39.9 kg/m2 BMI
* White/Caucasian
* Female
* Sedentary

Exclusion Criteria:

* Known cardiovascular, pulmonary, metabolic disease
* Pregnant females
* Any excluded criteria with MRI scans (i.e. certain metal implants, recent tattoos)
* Diabetic
* Hypertension
* Cigarette smoking
* MRI related contraindications (metal, no removable devices, etc.)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Changes in Visceral Abdominal Tissue (VAT) | 2 assessment periods: at baseline and week 4
  Changes in VAT will be measured using Magnetic Resonance Imaging

SECONDARY OUTCOMES:
Changes in Subcutaneous Abdominal Tissue (SAT) | 2 assessment periods: at baseline and week 4
  Changes in SAT will be measured using Magnetic Resonance Imaging
Changes in Muscular Strength | 2 assessment periods: at baseline and week 4
  Changes in muscular strength will be assessed by one-repetition maximum test on leg press and bench press
Changes in Cardiorespiratory Function | 2 assessment periods: at baseline and week 4
  Changes in cardiorespiratory will measured on a treadmill with a metabolic cart
Changes in fat mass (kg) | 2 assessment periods: at baseline and week 4
  Changes in fat mass will be measured using dual-energy x-ray absorptiometry
Changes in relative body fat (%BF) | 2 assessment periods: at baseline and week 4
  Changes in body composition (relative body fat, lean body mass and fat mass) will be measured using dual-energy x-ray absorptiometry
Changes in relative lean body mass (kg) | 2 assessment periods: at baseline and week 4
  Changes in lean body mass will be measured using dual-energy x-ray absorptiometry
Changes in Lipid profile (TG, Total Cholesterol, HDL2 HDL3, LDL) | 2 assessment periods: at baseline and week 4
  Samples will be processed to obtain serum and plasma, and stored at -80°c until analysis
Changes in concentration of Troponin | 2 assessment periods: at baseline and week 4
  Will be performed using a Luminex MAGPIX System with xPONENT 4.2
Changes in concentration of Fibrinogen | 2 assessment periods: at baseline and week 4
  Will be performed using a Luminex MAGPIX System with xPONENT 4.2
Changes in concentration of C-reactive protein (CRP) | 2 assessment periods: at baseline and week 4
  Will be performed using a Luminex MAGPIX System with xPONENT 4.2
Changes in concentration of IL-6 | 2 assessment periods: at baseline and week 4
  Will be performed using a Luminex MAGPIX System with xPONENT 4.2
Changes in concentration of IL-10 | 2 assessment periods: at baseline and week 4
  Will be performed using a Luminex MAGPIX System with xPONENT 4.2
Changes in concentration of TNF-alpha | 2 assessment periods: at baseline and week 4
  Will be performed using a Luminex MAGPIX System with xPONENT 4.2

CONTACTS AND LOCATIONS:
Overall Officials: Maria Fernandez del Valle, PhD, Principal Investigator — Southern Illinois University of Edwardsville
Locations (1):
- Southern Illinois University of Edwardsville, Edwardsville, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided